CLINICAL TRIAL: NCT03695120
Title: Renin Angiotensin Aldosterone Optimization in Acute Decompensated Heart Failure
Brief Title: RAAS Optimization for Acute CHF Patients
Acronym: ROAD-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201702923
Record Dates: First submitted 2018-09-19; First posted 2018-10-03 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Acute Decompensated Heart Failure
Keywords: ACEI (Angiotensin-Converting-Enzyme Inhibitor); ARB (Angiotensin II Receptor Blocker); CHF (Congestive Heart Failure); RAAS (Renin Angiotensin Aldosterone System)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The subjects will be randomized into a control group or variable group with an approximate 50/50 randomization. The control group will consist of subjects receiving ACEIs/ARBs. The variable group will consist of subjects that will not receive ACEI/ARBs during the first 72 hours of admission.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full Dose ACEI/ARB or Home Dose Group (No Intervention): This group will receive the full dose of ACEI/ARBs.
- No ACEI/ARB Group (Active Comparator): This group will not receive the full dose of ACEI/ARBs for the first 72 hours of hospitalization.
  Interventions: Other: Change of treatment plan

INTERVENTIONS:
Other: Change of treatment plan — Withholding ACEI/ARBs during initial 72 hours of admission with acute decompensated heart failure may help preserve renal function with a lesser decline in GFR. This treatment modification will also allow the option of aggressive diuresis in volume overloaded CHF patients which should result in a lesser decline of AKI, length of stay, readmission rates, and cost associated with CHF treatment.
  Arms: No ACEI/ARB Group

SUMMARY:
Holding ACEI/ARBs during initial 72 hours of admission with acute decompensated heart failure may help preserve renal function with a lesser decline in GFR. This treatment modification will also allow the option of aggressive diuresis in volume overloaded CHF patients which should result in a lesser decline of AKI, length of stay, readmission rates, and cost associated with CHF treatment.

DETAILED DESCRIPTION:
The investigators hypothesize that worsening renal function can be mitigated by withholding ACEI/ARB during the initial phase of in-patient treatment with aggressive diuresis. This hypothesis will be tested by randomly allocating 360 admitted patients with ADHF on two treatment paths: 1) no ACEI/ARB administered for initial 72 hours of treatment during aggressive diuresis versus 2) full dose ACEI/ARB administered concurrently with aggressive diuresis in naïve patients/home dose, who are already on such therapy. The study team hopes to find that holding ACEI/ARBs during the initial 72 hours of admission with acute decompensated systolic heart failure will help preserve renal function, as demonstrated by a lesser decline in GFR. In addition, this treatment would allow the option of aggressive diuresis in volume overloaded CHF patients, resulting in a lesser decline of AKI, length of stay, readmission rates, and costs associated with CHF treatment. By understanding the complex interaction between holding ACEIs/ARBs and continued aggressive diuresis, the investigators intend to develop optimal dosing strategies for acute, decompensated CHF patients, further minimizing adverse events such as electrolyte issues and declining GFR/AKI.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for enrollment if within the previous 24 hours they were treated with acute decompensated heart failure or diagnosed on the basis of the investigator's clinical diagnosis of heart failure, which needs to be supported by at least 2 the following criteria:

* Elevated concentration of B-type natriuretic peptide (BNP) or N-terminal pro-BNP. (Elevated BNP" defined as >300 for sinus rhythm, >500 for patients will atrial fibrillation and elevated pro BNP defined as >1000 for sinus rhythm, >1600 for atrial fibrillation.)
* Pulmonary edema on physical examination.
* Radiologic pulmonary congestion or edema.
* History of Chronic Heart Failure. Anticipated need for IV loop diuretics for at least 48 hours
* Willingness to provide informed consent

Exclusion Criteria:

* Previously diagnosed end-stage renal disease; Serum Potassium >5.5 mmol/L
* Cardiogenic Shock within 48 hours, ST-segment elevation myocardial infarction, ongoing ischemia.
* Need for renal replacement therapy through dialysis or ultrafiltration
* Myocardial infarction within 30 days of screening.
* Patients with systolic blood pressure of less than 90 mm Hg.
* Patients requiring Intravenous Vasodilators or inotropic agents (other than Digoxin) for heart failure
* BNP less than 250 ng/ml and/or proBNP less than 1000 mg/ml
* Pregnant women, prisoners, and institutionalized individuals
* Severe stenotic valvular disease
* Complex congenital heart disease
* Need for mechanical hemodynamic support
* Sepsis
* Terminal illness (other than HF) with expected survival of less than one year
* Previous adverse reaction to the study drugs
* Use of IV iodinated radiocontrast material in last 72 hours or planned during hospitalization
* Enrollment or planned enrollment in another randomized clinical trial during this hospitalization
* Inability to comply with planned study procedures
* Primary admission diagnosis other than acute heart failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Serum Creatinine Levels | Baseline, 24 hours, 48 hours, 72 hours
  Change in serum creatinine from randomization. (AKI is defined as an increase in the serum creatinine level of more than 0.3 mg per deciliter over 48 hours)
Patient Global Assessment (well-being) over 72 hours | 0 hours, 24 hours, 48 hours, 72 hours
  Patient global assessments by modified scale (based on Borg and VAS) for 0, 24, 48, 72 hours. Scaled 1 - 10. A "1" means the patient feels the best they've ever felt and a "10" means the participant feels the worst they have ever felt. Following all time points collected, the area under the curve for global assessment over the first 72 hours will be a primary efficacy endpoint (AUC for PGA).
  For patient well-being (PGA)
  1 Best I've ever felt 2 3 Feeling good 4 5 Feeling okay 6 7 Feeling bad 8 9 Feeling terrible 10 Worst I've ever felt
Dyspnea (shortness of breath) clinical change over 72 hours | 0 hours, 24 hours, 48 hours, 72 hours
  Patient dyspnea assessments by modified scale (based on Borg and VAS) for 0, 24, 48, 72 hours. Scaled 1 - 10. A "1" means no shortness of breath and a "10" means the patient can't breathe at all. Following all time points collected, the area under the curve for dyspnea assessment over the first 72 hours will be a primary efficacy endpoint (AUC for dyspnea).
  For shortness of breath (SOB)
  1 No SOB at all 2 3 Slight SOB 4 5 Moderate SOB 6 7 Severe SOB 8 9 Extreme SOB 10 "I can't breathe!"
Kinetic EGFR Levels | Baseline, 24 hours, 48 hours, 72 hours
  Change in kinetic EGFR from baseline to 24, 48, and 72 hours.

SECONDARY OUTCOMES:
Weight Change | Baseline, 24 hours, 48 hours, 72 hours
  Change in patient's weight over 3 day period.
Negative Fluid Balance | Baseline, 24 hours, 48 hours, 72 hours
  Changes in net fluid loss over 24, 48, 72 hours.
CHF Clinical Change | Baseline, 72 hours
  Change in signs and symptoms of congestion (defined as jugular venous pressure of <8 cm, with no orthopnea and with trace peripheral edema or no edema) from baseline to 24, 48, 72 hours.
Change in Renal Function | Baseline, 48 hours
  Renal biomarker (NephroCheck) levels at baseline and 48 hours. All patients receive baseline NephroCheck, and 48 hour re-assessment is limited to the first 100 patients.
Number of patients experiencing CHF Treatment Failure | Over 72 hours
  Persistent or worsening heart failure requiring additional interventions. Patients requiring other intravenous vasoactive medications for heart failure (inotropes, vasodilators, etc) for clinical reasons during the randomization period will meet the secondary endpoints of "worsening or persistent heart failure" and "treatment failure."
  Patients deemed to have a clinical need for additional diuretics during the study period will be permitted to receive diuretics. This will be captured as "rescue therapy" and will meet criteria for secondary endpoints of "worsening or persistent heart failure" and "treatment failure" endpoints.
  Conversely, patients may develop signs or symptoms of over-diuresis (such as hypotension) that will necessitate holding or discontinuing diuretics before completion of the randomization period. This will be captured as a "treatment failure" if it requires specific intervention beyond simply holding diuretics.
Hospitalization LOS | Total stay during current admission
  Length of inpatient stay
Cost Analysis | Total stay during current admission
  Cost of inpatient stay during admission.
Number of patient mortality | 30 days
  Death within 30 days of current inpatient stay (from first day of admission)
Number of patients readmitted or experiencing a ED visit | 30 days
  Readmission or ED visit at UF Health within 30 days of current inpatient stay (from first day of admission)
Number of patients readmitted over one year | 1 year
  Readmission at UF Health within 1 year of current inpatient stay (from first day of admission)

CONTACTS AND LOCATIONS:
Overall Officials: Bhagwan Dass, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Dass B, Dimza M, Singhania G, Schwartz C, George J, Bhatt A, Radhakrishnan N, Bansari A, Bozorgmehri S, Mohandas R. Renin-Angiotensin-Aldosterone System Optimization for Acute Decompensated Heart Failure Patients (ROAD-HF): Rationale and Design. Am J Cardiovasc Drugs. 2020 Aug;20(4):373-380. doi: 10.1007/s40256-019-00389-7. PMID 31797310